CLINICAL TRIAL: NCT03387826
Title: A Randomized, Pharmacodynamic Comparison of Low Dose Ticagrelor (60mg Bid) to Low Dose Prasugrel (5mg od) in Patients With Prior Myocardial Infarction
Brief Title: Low Dose Ticagrelor Versus Low Dose Prasugrel in Patients With Prior Myocardial Infarction
Acronym: ALTIC-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, National and Capodestrian University of Athens, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AttikonH14005
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Myocardial Infarction; Diabetes Mellitus; Coronary Artery Disease; Renal Disease
Keywords: ticagrelor; prasugrel
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus; Coronary Artery Disease; Kidney Diseases | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 60mg twice daily followed by Prasugrel 5mg once daily
  Interventions: Drug: Ticagrelor 60 mg; Drug: Prasugrel 5mg
- Prasugrel (Active Comparator): Prasugrel 5m once daily followed by Ticagrelor 60mg twice daily
  Interventions: Drug: Ticagrelor 60 mg; Drug: Prasugrel 5mg

INTERVENTIONS:
Drug: Ticagrelor 60 mg — Ticagrelor 60 mg twice daily
Drug: Prasugrel 5mg — Prasugrel 5 mg once daily

SUMMARY:
Taken together the results from DAPT and PEGASUS-TIMI54, it appears that physicians may consider extending beyond 1 year or reinitiating treatment with a thienopyridine or ticagrelor 60mg bid in patients with a prior MI and features of high ischemic and low bleeding risk. Comparative clinical or pharmacodynamic studies, however, between prasugrel 5 mg od and ticagrelor 60 mg bid in the chronic phase of stable post MI patients have not been performed.

In light of this, we believe that a dedicated pharmacodynamic study of ticagrelor 60 bid mg vs prasugrel 5 mg od in a PEGASUS-like population would be informative for the practicing clinician, thus setting the rationale for conducting this specifically designed investigation.

DETAILED DESCRIPTION:
This is a prospective, randomized, single blind, single center, crossover study. Eligible patients undergoing P2Y12 receptor antagonist therapy before screening will undergo a 14-day minimum washout period before randomization. Following screening/washout period (visit 1), patients will be randomized (visit 2, time 0) in 1:1 fashion to either prasugrel 5 mg od or ticagrelor 60 mg bid. Following 14±2 days (visit 3) patients will receive alternate treatment for additional 14 days (visit 4). Platelet reactivity assessment will be performed with the VerifyNow P2Y12 reaction assay at time 0, prior to first study drug dose. At visit 3 platelet function will be assessed at 2-4 hours post dose and prior to crossover. At visit 4 also platelet function will be assessed at 2-4 hours post study drug post dose. All patients will receive concomitant aspirin (100 mg/d) and standard secondary prevention medication.

The primary endpoint is the platelet reactivity measured in P2Y12 reaction units (PRU) at the end of the 2 study periods (pre-crossover and post-crossover).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Post-menopausal female (defined as absence of any vaginal bleeding for a year) or male aged >50 years
3. A spontaneous MI (ST or Non ST segment elevation) 1 to 3 years before enrolment. In addition, at least one of the following high-risk features: age of 65 years or older, diabetes mellitus requiring medication, a second prior spontaneous MI, multivessel coronary artery disease, or non-end stage renal disease (estimated creatinine clearance of <60 ml per minute).

Exclusion Criteria:

1. Planned use of a P2Y12 receptor antagonist, dipyridamole, cilostazol, or anticoagulant therapy during the study period;
2. Known allergy, intolerance, hypersensitivity to ticagrelor or prasugrel or any excipients,
3. Active pathological bleeding, severe hepatic impairment, a bleeding disorder or a history of an ischemic stroke or intracranial bleeding, a central nervous system tumor, or an intracranial vascular abnormality;
4. Gastrointestinal bleeding within the previous 6 months or major surgery within the previous 30 days;
5. Concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole, grapefruit juice over 1 litre daily), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine).
6. Increased risk of bradycardic events (e.g. known sick sinus syndrome or third degree AV block or previous documented syncope suspected to be due to bradycardia unless treated with a pacemaker).
7. Inability to adhere to the follow-up requirements or any other reason or condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity measured in P2Y12 reaction units (PRU) at the end of the 2 study periods | 14 days
  Platelet reactivity measured in P2Y12 reaction units (PRU) at the end of the 2 study periods (pre-crossover and post-crossover).

SECONDARY OUTCOMES:
High platelet reactivity rate at the end of the 2 study periods | 14 days
  High platelet reactivity rate (defined as >208 PRU) at the end of the 2 study periods
VerifyNow P2Y12 assay % inhibition, using the TRAP-induced response at the end of the 2 study periods | 14 days
  VerifyNow P2Y12 assay % inhibition, using the TRAP-induced (BASE channel) response at the end of the 2 study periods

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Alexopoulos, MD, Principal Investigator — Attikon Hospital
Locations (1):
- Attikon University Hospital, Chaïdári, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730